CLINICAL TRIAL: NCT06700174
Title: A Multicenter, Prospective, Single-arm, Observational Study
Brief Title: Lifetech AcuMark™ Sizing Balloon Post-Market Clinical Follow-up Study
Status: Recruiting | Type: Observational
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: LT/TS/571I-2023
Record Dates: First submitted 2024-11-15; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Atrial Septal Defect (ASD)
MeSH Terms: conditions — Heart Septal Defects, Atrial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
The objective of this PMCF study is to:

* confirm the safety and performance of the AcuMarkTM Sizing Balloon
* identify previously unknown side-effects
* monitor the identified side-effects (related to the procedure or to the medical devices)

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been confirmed with single secundum atrial septal defect (ASD) by echocardiography;
2. The anatomy of ASD is suitable for percutaneous closure;
3. Patients are scheduled to perform ASD closure;
4. Patients or legally authorized representative(s) who are willing and capable of providing informed consent.

Exclusion Criteria:

1. Any contraindication for ASD closure;
2. Patients have ostium primum ASD or coronary sinus ASD;
3. Patients who are pregnant or breastfeeding;
4. Patient is currently participating in another clinical trial that has not yet completed its primary endpoint.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with echocardiographic confirmation of a single secundum atrial septal defect (ASD) who are scheduled to undergo ASD closure.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Sizing success rate | At procedure
  The size of the selected occluder is proper by echocardiography observing
Incidence of major adverse events (MAEs) | From attempted procedure to discharge, up to 14 days
  Major adverse events are defined as stroke, occluder embolization, arrhythmia, thromboembolic event, oversizing of the defect, cardiac tamponade, and other procedure and/or device-related complications requiring re-intervention.

SECONDARY OUTCOMES:
Device success rate | At procedure
  Study device is successfully delivered in place and dilated without rupture and is successfully withdrew.
Incidence of procedure and/or device-related complications | From attempted procedure to discharge, up to 14 days
  Complications include vessel perforation/dissection, thromboembolism, hematoma, arrythmia, expansion of the defect, balloon migration, obstruction of venous return from the inferior vena cava.
Incidence of Serious Adverse Events | From attempted procedure to discharge, up to 14 days
Incidence of Device Deficiency (DD) | From attempted procedure to discharge, up to 14 days

CONTACTS AND LOCATIONS:
Locations (5):
- Turkey (Türkiye) (5):
  - Ankara (Bilkent) City Hospital, Ankara
  - Gazi Yasargil Woman and Child Hospital, Diyarbakır
  - Gaziantep University Hospital, Gaziantep
  - SiyamiErsek Thoracic and Cardiovascular Surgery Training and Research Hospital, Istanbul
  - Tepecik Training and Research Hospital, Izmir